CLINICAL TRIAL: NCT03374865
Title: Is the Medium the Message? A Study of the Affordances of Video-mediated Medical Consultations Compared to Traditional Consultations
Brief Title: Is the Medium the Message?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-2822
Record Dates: First submitted 2017-06-15; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-06

CONDITIONS: Video-mediated Consultation; Face to Face Consultation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Video-mediated consultation: Consultations using Facetalk videocommunication software
  Interventions: Other: Facetalk
- Face-to-face consultation: Traditional face-to-face consultations
  Interventions: Other: Face-to-face consultation

INTERVENTIONS:
Other: Facetalk — Area of interest: communication during Facetalk consultations
  Groups: Video-mediated consultation
Other: Face-to-face consultation — Area of interest: communication during face-to-face consultations
  Groups: Face-to-face consultation

SUMMARY:
Digital communication media like video-interaction (cf. Skype) are increasingly being adopted in institutional environments like hospitals for physician-patient interactions. We may expect that the use of a digital medium affects these interactions in various ways and on various levels. In video-interaction, eye contact for example is impossible due to the position of the camera, which implies interactional behavior through gaze is impaired. This may influence who speaks when, if and how the participants avoid/ solve misunderstandings, etcetera. This project makes headway in our understanding of the impact of new communication media on the role of language-in-use as a rich semiotic system, specifically in institutional interaction. This type of contextualized research reveals which communicative aspects users consider important, how they manage their institutional relationship through them and how they go about solving communication problems.

The project compares the interaction of physicians and patients in video-mediated consultations to their traditional, face-to-face counterparts on both the verbal and the nonverbal (gaze) level. The affordances of video-consultations with relevance to institutional goals and identities are analyzed through a comparison with the interaction in face-to-face consultations. The approach used is Conversation Analysis, which involves finding patterns on both the verbal and non-verbal level (in sequences, turn design, preference, etc.) in order to answer the question what goals and tasks the participants achieve and what dilemma's or problems they aim to solve in their talk. This study will provide insights in the limitations and advantages of both channels of communication. Best practices will be generated and outcomes of the analyses will be used to develop reco

DETAILED DESCRIPTION:
Research questions This project as a whole aims to understand the affordances of video-consultations. The general research question is: What are the interactional affordances of video-consultations compared to traditional consultations with respect to the goals and tasks the participants achieve and the dilemma's or problems the participants (aim to) solve in their talk?

Methodology The project involves a comparison of face-to-face and video-mediated consultations through the lens of affordances.

Data Baseline parameters, the Big Five survey, and details on experience and affinity with video consultation and (social) media use are obtained by means of a questionnaire. The patients are offered video-consultation as an option, so all video-consultation data involve patients with a certain level of openness and willingness towards the medium. The first set of data will consist of the recordings of 25 face-to-face and 25 videoconsultations of physicians with patients who have had a cancer resection, were discharged from the hospital and have a follow-up 'visit' in which the pathology results of the resection are reported. The reason for using video consultations for this group is that the patients would optimally benefit from not having to travel to the hospital, because the patients recently underwent surgery and are still recovering. These consultations solely consist of talk (no physical examination), so video consultation is possible here. Other medical departments have already implemented video consultations for similar reasons. All surgeons are in a similar stage of their career and the patients are recorded only once during follow-up consultation after surgery. The video-consultations are conducted through "Facetalk", video-interaction software. The physicians are trained to use this software and do about 3 to 4 videoconsultations per week. The face-to-face consultations are recorded with two camera's. The video-interaction data consist of recordings of the physician's screen during the consultation and a video-recording of the physician in the physical environment (sitting at a desk), capturing the physician's body and head movement to and away from the video-interaction screen (e.g., towards a second computer screen with the patient's file). The main applicant is already acquainted with the setting through the observation of video-consultations from within the physician's office.

In addition to the video-recordings, brief surveys will be conducted with patients and physicians after the consultation to measure satisfaction with the consultation. Informed consent for the study and related education will be sought from both the patients and the surgeons. The participants will also be asked for permission to archive the videorecordings for future research on authentic communication. The recordings will be stored in a safe at the Centre for Language Studies, Radboud University. Single episodes will be saved occasionally on the researchers' computer for the benefit of the study (data session). These episodes will be removed again as soon as possible. The participants will be anonymized in the transcripts and any publication and conference presentation that may follow from this study. Anonymization is achieved through functionalities in Windows Movie Maker (drawing effect) and Audacity (tone adaptation). Rendering participant unrecognizable means that the audience (of a presentation/ readers of an article) would not be able to recognize participants without prior knowledge of the hospital, the department etc. These adaptations do not affect the value of the material because non-verbal behavior (head shakes, gestures) and the talk are still understandable in combination. It is acceptable and common in the academic domain that recordings shown at conferences and in publications are anonymized.

Before the patient is resigned from the hospital after surgery, the surgeon will ask the patient whether the patient prefers a f2f or video consultation. Then, the patient will be asked by the doctor whether the patient gives permission to be approached for participation in the study. If yes, the patient information will be mailed to the patient to read and consider at home. Permission (including signature) can be e-mailed to the researcher or given to the doctor in person prior to the consultation. After that, the doctor will also give permission and sign. It is possible at any time for the participants to withdraw from the study and have the video consultation interrupted. To withdraw from the study they should e-mail the main researcher of the project. This is explained in the patient information.

Method The analysis will be qualitative (micoanalytic) and iterative. The main method is multimodal conversation analysis. Conversation analysis has a long tradition of research based on the rendition of talk and interaction in terms of written transcripts of the audible cues. The video mediated and face-to-face interactions will be compared. This means that phenomena observed in the video-mediated consultations will be compared to equivalent actions and practices in the face-to-face consultations, both verbal and non-verbal. Relevant phenomena are likely to be the opening of the conversation (checking the technology), the design of questions (use of more lexical tokens than deixis), particular gestures, specific repair sequences due to technical trouble etc.). The analysis will be descriptive and will result in recommendations for doing videoconsulting.

All talk will be transcribed according to CA conventions . Software like ELAN may be used for the synchronization of multiple video data and for the annotation of (fragments of) the video data.

ELIGIBILITY:
Inclusion Criteria:

* Discharged post-operative patients
* Follow up consultation for pathology results

Exclusion Criteria:

- Physical examination needed

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Discharged post-operative patients from a single tertiary medical center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Verbal communication | 10 minutes
  Verbal communication. The main method is multimodal conversation analysis. Conversation analysis has a long tradition of research based on the rendition of talk and interaction in terms of written transcripts of the audible cues. The video-mediated and face-to-face interactions will be compared. This means that phenomena observed in the video-mediated consultations will be compared to equivalent actions and practices in the face-to-face consultations. Relevant phenomena are likely to be the opening of the conversation (checking the technology), the design of questions (use of more lexical tokens than deixis), particular gestures, specific repair sequences due to technical trouble etc.). The analysis will be descriptive.
  All talk will be transcribed according to CA conventions. Software like ELAN may be used for the synchronization of multiple video data and for the annotation of (fragments of) the video data.

SECONDARY OUTCOMES:
Non-verbal communication | 10 minutes
  Body language

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No